CLINICAL TRIAL: NCT05204368
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Comparative, Phase 3 Study to Evaluate the Efficacy and Safety of Intravenous Imipenem/Cilastatin/XNW4107 in Comparison With Meropenem in Hospitalized Adults With Complicated Urinary Tract Infections, Including Acute Pyelonephritis.(EudraCT no. 2022-000061-40)
Brief Title: Evaluation of the Efficacy and Safety of Intravenous Imipenem/Cilastatin/XNW4107 in Comparison With Meropenem in Hospitalized Adults With cUTI Including AP (EudraCT no. 2022-000061-40)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XNW4107-301
Record Dates: First submitted 2022-01-05; First posted 2022-01-24 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Complicated Urinary Tract Infection Including Acute Pyelonephritis
MeSH Terms: interventions — Cilastatin; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Imipenem/Cilastatin/XNW4107 (Experimental): Imipenem/Cilastatin 500mg/500mg in combination with XNW4107 250mg ,q6h(0.5h infusion)
  Interventions: Drug: Combination of Imipenem/Cilastatin and XNW4107
- Meropenem (Active Comparator): Meropenem 1g ,q8h (0.5h infusion)
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Combination of Imipenem/Cilastatin and XNW4107 — Imipenem/Cilastatin 500mg/500mg and XNW4107 250mg for injection
  Arms: Imipenem/Cilastatin/XNW4107
Drug: Meropenem — Meropenem 1g for injection
  Arms: Meropenem

SUMMARY:
This is A Multicenter, Randomized, Double-Blind, Double-Dummy, Comparative, Phase 3 Study to Evaluate the Efficacy and Safety of Intravenous Imipenem/Cilastatin/Funobactam in Comparison with Meropenem in Hospitalized Adults with Complicated Urinary Tract Infections, including Acute Pyelonephritis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing and able to provide written informed consent.
2. Willing and able to comply with all study assessments and adhere to the protocol schedule.
3. Hospitalized or requiring hospitalization for cUTI or AP in male or female patients ≥18 years on the day of signing informed consent.
4. Requiring treatment with IV antibiotic therapy.
5. Evidence of AP or cUTI

   At least 1 of the following:
   * Nausea or vomiting.
   * Chills or rigors or warmth associated with fever (temperature >38°C).
   * Peripheral white blood cell count (WBC) >10,000/mm³ or bandemia , regardless of WBC count.
6. Having at least 1 of the following complicated factors for cUTI (not required for AP):

   1. Indwelling catheter of the urinary tract.
   2. Urinary retention.
   3. Any functional or anatomical abnormality of the urogenital tract resulting in at least 100 mL or more of residual urine after voiding.
   4. Obstructive uropathy .
7. Evidence of pyuria demonstrated by 1 of the following methods:

   1. Dipstick analysis positive for leukocyte esterase.
   2. ≥10 WBCs per µL in unspun urine, or ≥10 WBCs per high power field in spun urine.

Exclusion Criteria:

1. Patients with any of the following conditions:

   1. Suspected or confirmed perinephric abscess
   2. Suspected or confirmed renal corticomedullary abscess
   3. Suspected or confirmed acute or chronic bacterial prostatitis, orchitis, or epididymitis, as determined by history and/or physical examination
   4. Known polycystic kidney disease or only 1 functional kidney
   5. Known chronic vesicoureteral reflux
   6. Previous renal transplantation or planned renal transplantation within 2 weeks of study entry
   7. Patients receiving renal replacement therapy
   8. Complete, permanent obstruction of the urinary tract
   9. Urinary tract symptoms attributable to a sexually transmitted disease.
2. Gross hematuria requiring intervention other than administration of study drug.
3. Urinary tract surgery within 7 days prior to randomization or urinary tract surgery planned during the study period (except surgery required to relieve an obstruction or place a stent or nephrostomy).
4. Patient has any urinary catheter or device that will not be removed or replaced (if removal is not clinically acceptable) during IV therapy, including but NOT limited to indwelling bladder catheters, ureteral catheters, suprapubic catheters, J stents, and nephrostomy tubes.
5. Renal function at Screening as estimated glomerular filtrated rate <15 mL/min/1.73㎡, calculated using Modification of Diet in Renal Disease.
6. Known non-urinary tract source of infection such as endocarditis, osteomyelitis, abscess, meningitis, or pneumonia diagnosed within 7 days prior to randomization.
7. Any rapidly progressing disease or immediately life-threatening illness, including, but not limited to, current or impending respiratory failure, septic shock, acute heart failure, acute coronary syndrome, unstable arrhythmias, hypertensive emergency, acute hepatic failure, active gastrointestinal bleeding, profound metabolic abnormalities (e.g., diabetic ketoacidosis), or acute cerebrovascular events.
8. If the culture result is available prior to randomization and identifies only a Gram-positive pathogen and/or only a Gram negative pathogen (>10^5 CFU/mL) known to be resistant to meropenem
9. If the culture result is available prior to randomization and identifies isolates >2 pathogens or no pathogens with >10^5 CFU/mL identified or patient has a confirmed fungal UTI.
10. Receipt of more than 24 hours of a potentially effective systemic antibacterials within 72 hours prior to start of study therapy.
11. History of a seizure disorder.
12. Female patients of childbearing potential, who are unable or unwilling to use a highly effective method of birth control during the study and for at least 30 days following the last dose of study medication.
13. A female who is pregnant or breastfeeding, or have a positive pregnancy test at Screening.
14. Patient is participating in any clinical study of any investigational medication (i.e., non-licensed medication) during the 30 days prior to randomization. COVID-19 vaccines that are given under emergency use authorization are not considered investigational agents.
15. Documented presence of immunodeficiency or an immunocompromised condition including hematologic malignancy, bone marrow transplant, known human immunodeficiency virus infection with a CD4 count <200/mm³, or requiring frequent or prolonged use of systemic corticosteroids or other immunosuppressive drugs.
16. Patients with 1 or more of the following laboratory abnormalities in baseline specimens: aspartate aminotransferase, alanine aminotransferase >3 × the upper limit of normal (ULN), total bilirubin level >2 × ULN (except for isolated hyperbilirubinemia due to known Gilbert's disease), neutrophils <500 cells/mm³, platelet count <40,000/mm³
17. Patients requires concomitant medication with valproic acid or divalproex.
18. History of active liver disease, cirrhosis.
19. Documented or severe hypersensitivity or previous severe adverse drug reaction, especially to any beta-lactam antibiotics, or any of the excipients used in the study drug formulations.
20. Any other condition or prior therapy, which, in the opinion of the investigator, would make the patient unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
overall success | Day 21[±2 days]
  The proportion of patients who achieve overall success at the Test of cure(TOC) visit in the micro-modified-intent-to-treat(micro-MITT) population.
  Overall success requires symptomatic clinical success and microbiologic success at the TOC visit.

SECONDARY OUTCOMES:
overall success | EOT: from treatment day 7 up to day 15
  The proportion of patients who achieve overall success at the End of treatment (EOT) visit in the micro-MITT population.
overall success | Day 28[±3 days]
  The proportion of patients who achieve overall success at the Late follow-up(LFU) visit in the micro-MITT, extended micro-MITT, Clinically evaluable(CE), Microbiologically evaluable(ME) populations.
symptomatic clinical success | Day 4; EOT: from treatment day 7 up to day 15; TOC: Day 21[±2 days]; LFU: Day 28[±3 days]
  The proportion of patients with symptomatic clinical success at Day 4, EOT, TOC, and LFU visit in the micro-MITT, extended micro-MITT, CE, and ME populations
microbiological success | EOT: from treatment day 7 up to day 15; TOC: Day 21[±2 days]; LFU: Day 28[±3 days]
  The proportion of patients with microbiological success at EOT, TOC, and LFU visit in the micro-MITT, extended micro-MITT, and ME populations
By-pathogen microbiological success | EOT: from treatment day 7 up to day 15; TOC: Day 21[±2 days]; LFU: Day 28[±3 days]
  The proportion of patients with by-pathogen microbiological success at EOT, TOC, and LFU visit in the micro-MITT, extended micro-MITT, and ME populations
The proportion of overall success; symptomatic clinical, and microbiologic success | EOT: from treatment day 7 up to day 15; TOC: Day 21[±2 days]; LFU: Day 28[±3 days]
  The proportion of overall success; symptomatic clinical, and microbiologic success at EOT, TOC, and LFU visit in the Carbapenem-resistant-MITT(CR-MITT) population
clinical success | Day 21[±2 days]
  The proportion of patients with clinical success based on the investigator's assessment of clinical response at TOC visit in the micro-MITT population

CONTACTS AND LOCATIONS:
Overall Officials: Jason Le, Study Chair — Evopoint Biosciences Inc.
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States